CLINICAL TRIAL: NCT05712278
Title: A Phase I, Single-arm, Open Label, Dose Escalation, Multicenter Study of Off-the-shelf Natural Killer (NK) Cells (SAR445419) in Participants With Relapsed or Refractory Acute Myeloid Leukemia (R/R AML)
Brief Title: A Study to Investigate Use of Off-the-shelf Natural Killer (NK) Cells (SAR445419) in Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED17749; U1111-1279-2948 (Other: ICTRP)
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; fludarabine phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR445419 (Experimental): Treatment consists of chemotherapy with fludarabine 30mg/m2/day and cytarabine 2g/m2/day administered for 5 days (Day -6 to Day -2), followed by 6 doses of SAR445419 given thrice weekly for 2 weeks beginning Day 1.
  Interventions: Drug: SAR445419; Drug: fludarabine; Drug: cytarabine

INTERVENTIONS:
Drug: SAR445419 — Cell suspension, by intraveneous (IV) injection
Drug: fludarabine — Solution for injection , by IV injection
  Other Names: fludara
Drug: cytarabine — Solution for injection, by IV injection
  Other Names: cytosar-U

SUMMARY:
This is a single group, Phase 1, single-arm, dose escalation study to determine the candidate dose(s), and evaluate safety, tolerability, and preliminary anti-tumor activity of SAR445419 administered after fludarabine and cytarabine conditioning for the treatment of relapsed or refractory acute myeloid leukemia (R/R AML). Adult participants with R/R AML will be eligible for treatment.

The study is intended to assess the candidate dose(s) by the occurrence of dose-limiting toxicity (DLT) from start of chemotherapy until 28 days after the first administration of SAR445419.

The duration of the study for a participant will include:

* Screening period up to 21 days prior to initiating chemotherapy,
* Treatment period of 5 days chemotherapy followed by SAR445419 administered for 2 weeks and end of treatment visit 56 days after first SAR445419 administration,
* Survival follow-up period up to 1 year after the last participant has started treatment with SAR445419.

DETAILED DESCRIPTION:
Participants will be followed for 28 days (for DLT evaluations) after administration of the first SAR445419 dose (Day 1) for the primary endpoint and for 1 year after the first SAR445419 dose for selected secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Participant must be 18 years of age inclusive

Participants with confirmed diagnosis of relapsed or primary refractory acute myeloid leukemia (AML), according to World Health Organization (WHO) classification, including:

* Participants with relapsed AML after allogeneic stem cells transplantation, including those who have received donor lymphocyte infusions,
* Isolated central nervous system (CNS) or extramedullary disease,
* At least 1 prior line of therapy which includes chemotherapy, hypomethylating agents, venetoclax or targeted therapy.

Participants with a weight ≥42 kg.

Exclusion Criteria:

* Second primary malignancy that requires active therapy. Adjuvant hormonal therapy is allowed.
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or human immunodeficiency virus (HIV) disease requiring antiretroviral treatment, or having active hepatitis B or C infection, or symptomatic severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Pregnant or breast-feeding women, female participants of childbearing potential, and male participants with female partners of childbearing potential who are not willing to avoid pregnancy by using a highly effective method of contraception (2 barrier method or 1 barrier method with a spermicide, intrauterine device, or hormonal contraception with inhibition of ovulation, for 2 weeks prior to the first dose of SAR445419, during treatment, and 6 months after the last dose of fludarabine). A woman is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile.
* History of solid organ transplant, including corneal transplant.
* Receiving at the time of first SAR445419 administration corticosteroid as a concomitant medication with corticosteroid dose >10 mg/day of oral prednisone or the equivalent, except steroid inhaler, nasal spray, or ophthalmic solution
* Known contraindication to any of the non-investigational medicinal products (NIMPs) (fludarabine, cytarabine, acetaminophen and diphenhydramine).
* Concurrent treatment with other investigational drugs

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting (DLT) toxicity | from Day 1 to Day 28
Incidence of DLT from start of chemotherapy | From Day -6 to Day 28

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From baseline up to 1 year
Median time to neutrophil and platelet count recovery | From Day -6 up to 1 year
  Median time to neutrophil and platelet count recovery post chemotherapy
Rate of HSCT | From baseline up to 1 year
  Percentage of participants going onto hematopoietic stem cell transplantation (HSCT) following SAR445419 treatment but prior to subsequent therapy for treatment of AML
Number of participants with infection | From baseline up to 1 year
Number of participants by type of infection | From baseline up to 1 year
  Fungal, bacterial, viral, and particularly cytomegalovirus (CMV) infection or reactivation (opportunistic) infection
Percentage of participants with Composite Complete Remission (CRc) rate | From baseline up to Day 56
  Percentage of participants who have a complete remission (CR) or a complete remission with incomplete hematological recovery (CRi) as defined by the modified European LeukemiaNet (ELN) 2022 criteria for AML
Percentage of participants with alternative complete remission rate | From baseline up to Day 56
  Percentage of participants with CR or a complete remission with partial hematological recovery (CRh)
Percentage of participants with overall complete remission rate | From baseline up to Day 56
  Percentage of participants with CR or CRh or CRi or morphological leukemia-free state (MLFS)
Duration of response | From baseline up to 1 year
  Time interval from first documented evidence of CR until progressive disease (PD) as per modified ELN 2022 criteria for AML or death due to any cause, whichever comes first
Duration of event-free survival | From baseline up to 1 year
  Time interval from date of first SAR445419 administration to induction failure, relapse or death due to any cause, whichever comes first
Overall survival rate at 6 months | From baseline up to 6 months
  Time from the first SAR445419 administration to death from any cause
Overall survival rate at 1 year | From baseline up to 1 year
  Time from the first SAR445419 administration to death from any cause
Time to treatment failure | From baseline up to 1 year
  Time from first SAR445419 administration to discontinuation for any reason excluding remission

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - University of Nebraska Medical Center Site Number : 8400003, Omaha, Nebraska
  - Albert Einstein College of Medicine Site Number : 8400001, The Bronx, New York
  - ~MD Anderson Cancer Center Site Number : 8400002, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TED17749 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25362&tenant=MT_SNY_9011